CLINICAL TRIAL: NCT03698136
Title: Electrical Stimulation in Denervated Muscles of the Upper Limbs - Effect on Muscle Morphological Properties - a Pilot Study
Brief Title: Electrical Stimulation in Denervated Muscles of the Upper Limbs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-20
Record Dates: First submitted 2018-10-01; First posted 2018-10-05 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2021-05

CONDITIONS: Tetraplegia
Keywords: tetraplegia; denervated muscles; electrical stimulation
MeSH Terms: conditions — Quadriplegia

STUDY DESIGN:
Intervention Model Description: Repeated measurement interventional Single Subject Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stimulation of denervated muscle (Experimental): direct muscle stimulation 5 times a week for 33 minutes 3 minutes warm up 30 minutes treatment
  Interventions: Other: Stimulation of denervated muscles

INTERVENTIONS:
Other: Stimulation of denervated muscles — The study investigates the effect of electrical stimulation on denervated muscles in the forearm and hand regarding muscle structure and thickness. The study will be performed on tetraplegics who have either paralysed the wrist extensor, the short thumb spreader or the muscle between the thumb and index finger.The study lasts 12 weeks and consists of an ultrasound examination at the beginning and end of the study and an intermediate stimulation phase.The stimulation takes place either during an inpatient stay or at home for 12 weeks, 5 times a week 33 minutes.

SUMMARY:
In the last decade the stimulation of denervated muscles got more attention. Not at least because of the promising results of the RISE project (Use of electrical stimulation to restore standing in paraplegics with long-term denervated degenerated muscles). In this European project it was shown that electrical stimulation of denervated muscles in spinal cord injuries (SCI) increased muscle mass and improved the trophic situation of the lower extremities. Furthermore, structural altered muscle into fat- and connective tissue could be restored into contractile muscle tissue by stimulation. However, only a few studies investigated the effect of direct muscle stimulation in case of peripheral nerve damage in the upper extremities. None investigated the stimulation effect in denervated or partially denervated muscles in the upper extremities in tetraplegic patients.

DETAILED DESCRIPTION:
In the last decade the stimulation of denervated muscles became part of the rehabilitation of spinal cord injuries (SCI). Not at least because of the promising results of the RISE project (Use of electrical stimulation to restore standing in paraplegics with long-term denervated degenerated muscles). In this European project it was shown that electrical stimulation of denervated muscles in SCI increased muscle mass and improved the trophic situation of the lower extremities. Furthermore, structural altered muscle into fat- and connective tissue could be restored into contractile muscle tissue by stimulation. However it has been shown that an extended time after SCI hinders the stimulation impact. The denervation process can be divided in four chronologically running steps. Muscle fibrillations are present some days after lesion followed by a loss of tension during electrical evoked tetanic contraction. After months a severe disorganization of the contractile structure in the muscle occurs and finally ends after years in a replacement of muscle fibers into fat tissue and collagen. The best results have been seen within three years after SCI. A stimulation protocol should be set up to start with single twitches combined with tetanic stimulation patterns according to the patients' improvements. The progression in stimulation training to elicit a tetanic contraction - 40 ms pulse duration with a pulse pause of 10 ms and bursts of 2 sec - could last some month in chronic stage after SCI. The stimulation of denervated muscles of the upper extremities gets more attention. It has been investigated that the cross sectional area of denervated muscle fibers could have been increased by early electrical stimulation. Furthermore, the changes in myosin heavy chain isoform, following denervation could be reversed. That indicates that early onset of stimulation could preserve the contractile muscle structure for possible reinnervation or further treatment options. Specially for tetraplegic patients who could benefit from nerve transfers, could win time for their decision.

ELIGIBILITY:
Inclusion Criteria:

* traumatic or non-traumatic spinal cord injury
* acute and subacute (≥ 6 weeks) and chronic (≥ 2 years) spinal cord injury
* Age ≥ 18 years
* Level of lesion C3 - Th1
* American Spinal Injury Association Impairment Score (AIS) A/B/C/D
* denervated M. extensor carpi ulnaris or M. abductor pollicis brevis or M. interosseus
* Signed informed consent

Exclusion Criteria:

* innervated or partially innervated M. extensor carpi ulnaris or M. abductor pollicis brevis or M. interosseus
* Patients' inability to follow the study, e.g. mental-health problems, language problems, dementia etc.
* Pregnancy (anamnestic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Pennation angle (degrees) | Baseline and after 12 weeks of electrical stimulation
  Difference between the pennation angle of the stimulated muscle at baseline and after the stimulation period

SECONDARY OUTCOMES:
Muscle thickness (mm) | Baseline
  Muscle thickness at baseline
Questionaire on participant perception | after 12 weeks of electrical stimulation
  Participant perception of the treatment effectiveness scale to evaluate the feasibility of the treatment expenditure according to the benefit of the stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Jan Fridén, Prof.Dr.med., Principal Investigator — Swiss Paraplegic Research, Nottwil
Locations (1):
- Swiss Paraplegic Centre Nottwil, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bersch I, Koch-Borner S, Friden J. Electrical stimulation-a mapping system for hand dysfunction in tetraplegia. Spinal Cord. 2018 May;56(5):516-522. doi: 10.1038/s41393-017-0042-2. Epub 2018 Jan 22. PMID 29358674
- [Background] Modlin M, Forstner C, Hofer C, Mayr W, Richter W, Carraro U, Protasi F, Kern H. Electrical stimulation of denervated muscles: first results of a clinical study. Artif Organs. 2005 Mar;29(3):203-6. doi: 10.1111/j.1525-1594.2005.29035.x. PMID 15725217
- [Background] Helgason T, Gargiulo P, Johannesdottir F, Ingvarsson P, Knutsdottir S, Gudmundsdottir V, Yngvason S. Monitoring muscle growth and tissue changes induced by electrical stimulation of denervated degenerated muscles with CT and stereolithographic 3D modeling. Artif Organs. 2005 Jun;29(6):440-3. doi: 10.1111/j.1525-1594.2005.29073.x. PMID 15926978
- [Background] Gordon T, English AW. Strategies to promote peripheral nerve regeneration: electrical stimulation and/or exercise. Eur J Neurosci. 2016 Feb;43(3):336-50. doi: 10.1111/ejn.13005. Epub 2015 Aug 14. PMID 26121368
- [Background] Kern H, Boncompagni S, Rossini K, Mayr W, Fano G, Zanin ME, Podhorska-Okolow M, Protasi F, Carraro U. Long-term denervation in humans causes degeneration of both contractile and excitation-contraction coupling apparatus, which is reversible by functional electrical stimulation (FES): a role for myofiber regeneration? J Neuropathol Exp Neurol. 2004 Sep;63(9):919-31. doi: 10.1093/jnen/63.9.919. PMID 15453091